CLINICAL TRIAL: NCT06344702
Title: The Effect of Continuous Positive Airway Pressure Ventilation on Maternal and Infant Outcomes in Pregnant Women With Obstructive Sleep Apnea Syndrome
Brief Title: The Effect of CPAP on Maternal and Infant Outcomes in Pregnant Women With OSAS
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Guoli Liu, Chief Physician, Peking University People's Hospital
Other Study IDs: 2024PHB065-001
Record Dates: First submitted 2024-03-17; First posted 2024-04-03 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Maternal Hypertension
Keywords: gestational hypertension
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- The CPAP treatment group: CPAP standardized treatment+standard obstetric care
  Interventions: Device: CPAP
- OSAS control group: standard obstetric care
- Non OSAS group: standard obstetric care

INTERVENTIONS:
Device: CPAP — 70% of nights use CPAP for more than 4 hours
  Groups: The CPAP treatment group

SUMMARY:
The goal of this clinical trial is to learn about the impact of CPAP on the maternal and infant outcomes of women with obstructive sleep apnea syndrome. The main questions aim to answer are:

[question 1]Explore the impact of different CPAP treatment times on the maternal and infant outcomes of pregnant women with combined OSAS; [question 2]Explore the effects of CPAP on placental weight and birth weight/placental weight ratio in OSAS pregnant women.

The CPAP treatment group received standardized CPAP treatment and routine prenatal care, while the non CPAP treatment group and non OSAS group only received routine prenatal care.

DETAILED DESCRIPTION:
Selecting high-risk OSAS pregnant women who underwent sleep breathing monitoring at 24-28 weeks of pregnancy and were registered in the Obstetrics and Gynecology Department of Peking University People's Hospital from January 2024 to December 2025 as the study subjects, collecting baseline data, following up on the study subjects until delivery, collecting CPAP treatment time, maternal and infant outcome related indicators, and placental weight. Assessing high-risk factors for OSAS during prenatal checkups for pregnant women: symptoms, signs, clue diseases, Epworth scale; Select pregnant women who meet the high-risk factors for OSAS at 24-28 weeks and collect their baseline data and ESS scores; Sleep breathing tests were performed on high-risk OSAS pregnant women aged 24-28 weeks, and their AHI, ODI, and SaO2 were recorded; Set AHI ≥ 5 times/h as the OSAS group, with those receiving standard CPAP treatment being the CPAP treatment group, those refusing CPAP treatment being the non CPAP treatment group, and AHI<5 times/h as the non OSAS group. The CPAP treatment group received standardized CPAP treatment and routine prenatal care, while the non CPAP treatment group and non OSAS group only received routine prenatal care; Follow up the above research subjects until the end of delivery, collect their ESS scores, CPAP treatment time, maternal and infant outcome indicators, and placental weight after treatment. After trimming the fetal membrane and umbilical cord, weigh and measure the placenta. Use statistical methods to analyze baseline data and ESS scores before and after delivery; Analyze the outcomes of pregnant women in different CPAP treatment and control groups, including delivery methods, postpartum hemorrhage, and admission to the intensive care unit (ICU); The neonatal outcomes include gestational age, preterm birth, birth weight of the newborn, infants under gestational age, and umbilical artery blood gas analysis (pH<7.10, LAC>=6.0mmol/L, BE<-12mmol/L); Analyze the placental weight and birth weight/placental weight ratio in the CPAP treatment group, control group, and non OSAS group.

ELIGIBILITY:
Inclusion Criteria:

* (1)Pregnant women at 24-28 weeks of gestation
* (2)Apnea hypopnea index (AHI) AHI ≥ 5 times/h

Exclusion Criteria:

* (1)Multiple pregnancies or fetal malformations
* (2)Severe mental illness
* (3)Severe heart and lung disease or liver and kidney disease
* (4)Previous diagnosis of OSAS
* (5)Other sleep disorders

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The CPAP treatment group received CPAP standard treatment+standard obstetric care, while the OSAS control group and non OSAS group only received standard obstetric care. The effects of the two different treatment plans were observed.
Sampling Method: Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Explore the effects of CPAP on placental weight and birth weight/placental weight ratio in OSAS pregnant women. | April 1, 2024 to December 31, 2025
  Analyze the placental weight and birth weight/placental weight ratio in the CPAP treatment group, control group, and non OSAS group.

IPD SHARING:
Plan to Share IPD: Undecided